CLINICAL TRIAL: NCT02374307
Title: Effect of a Falls-prevention Exercise Program on Health-related Quality of Life in Older Fallers Receiving Home Care. A Randomized Controlled Trial
Brief Title: Falls Prevention in Older Home Care Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Maria Bjerk, PhD Research Fellow, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 130140; 2014/2051 (Other: Regional Ethics Committees Norway)
Record Dates: First submitted 2015-02-16; First posted 2015-02-27 (Estimated); Results first posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Accidental Falls
Keywords: Falls; Home care; Older people; Falls prevention; Quality of life; Exercise; Balance; Preventative care; Community health services; Home-help services
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and education (Experimental): This group performs a 12-week individual tailored home exercise programme in accordance with the manual of Otago exercise programme. Physiotherapists visit the participants 5 times during the 12 weeks (at week 1,2,4,8 and 10) to prescribe and progress exercises. Motivational conversations on telephone are performed the weeks when no visits are scheduled. Additionally, the participants receive information on the first visit which will focus on motivation, importance of adherence and effectiveness of falls prevention. The participants are expected to do exercises on their own, and in that way perform exercises 3 times weekly. If safe, the participant are provided with a walking plan and be encouraged to walk twice weekly.
  Interventions: Other: Exercise and education
- Control (No Intervention): The control group performs activities as usual.

INTERVENTIONS:
Other: Exercise and education — Exercise according to the falls prevention programme. Information on motivation, the effectiveness of falls prevention and the importance of adherence.
  Arms: Exercise and education

SUMMARY:
The aim of this study is to investigate the effect of a falls-prevention exercise programme on health-related quality of life, fear of falling, falls and physical function in older people receiving home care. Participants in the intervention group perform the Otago exercise programme. Participants in the control group continue their usual activities.

DETAILED DESCRIPTION:
Falls and falls-related injuries are considered a serious public health issue in the older population. Strength and balance exercise in combination with information about falls prevention seems to be effective in reducing falls, but less is known about the effect of this kind of intervention on quality of life. This randomized controlled trial investigates the effect of a falls prevention program on health-related quality of life, fear of falling, falls and physical function in community-dwelling older people who receive home care.

ELIGIBILITY:
Inclusion Criteria:

* has fallen at least one time in the last 12 months
* receives home-help services
* able to walk independently indoors with or without walking aid

Exclusion Criteria:

* medical contraindication to exercise
* life expectancy <1 year
* scores under 23 points on Mini Mental Scale Examination
* participating in another falls prevention programme during the 12 weeks of the programme, for example a falls prevention group

Min Age: 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 155 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Bergland, PhD, Study Director — OsloMet - Oslo Metropolitan University; Maria Bjerk, MSc, Principal Investigator — OsloMet - Oslo Metropolitan University
Locations (6):
- Norway (6):
  - Municipality of Frogn, Drøbak, Akershus
  - Municipality of Rælingen, Fjerdingby, Akershus
  - Municipality of Skedsmo, Lillestrøm, Akershus
  - Municipality of Lørenskog, Lørenskog, Akershus
  - Municipality of Bærum, Sandvika, Akershus
  - Municipality of Sørum, Sørumsand, Akershus

IPD SHARING:
Plan to Share IPD: No
The raw data collected in this project is only available to the participating researchers due to risk to confidentiality of participants and Norwegian data protection laws. An anonymized subset of the raw data, where direct and potentially indirect person identifiers are removed, is planned to be made available in a public data repository after the project is finished and main results are published.

REFERENCES:
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Brooks R. EuroQol: the current state of play. Health Policy. 1996 Jul;37(1):53-72. doi: 10.1016/0168-8510(96)00822-6. PMID 10158943
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Janssen MF, Pickard AS, Golicki D, Gudex C, Niewada M, Scalone L, Swinburn P, Busschbach J. Measurement properties of the EQ-5D-5L compared to the EQ-5D-3L across eight patient groups: a multi-country study. Qual Life Res. 2013 Sep;22(7):1717-27. doi: 10.1007/s11136-012-0322-4. Epub 2012 Nov 25. PMID 23184421
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Yardley L, Beyer N, Hauer K, Kempen G, Piot-Ziegler C, Todd C. Development and initial validation of the Falls Efficacy Scale-International (FES-I). Age Ageing. 2005 Nov;34(6):614-9. doi: 10.1093/ageing/afi196. PMID 16267188
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Vellas B, Guigoz Y, Garry PJ, Nourhashemi F, Bennahum D, Lauque S, Albarede JL. The Mini Nutritional Assessment (MNA) and its use in grading the nutritional state of elderly patients. Nutrition. 1999 Feb;15(2):116-22. doi: 10.1016/s0899-9007(98)00171-3. PMID 9990575
- [Background] Thomas S, Mackintosh S, Halbert J. Does the 'Otago exercise programme' reduce mortality and falls in older adults?: a systematic review and meta-analysis. Age Ageing. 2010 Nov;39(6):681-7. doi: 10.1093/ageing/afq102. Epub 2010 Sep 4. PMID 20817938
- [Background] Muir SW, Berg K, Chesworth B, Speechley M. Use of the Berg Balance Scale for predicting multiple falls in community-dwelling elderly people: a prospective study. Phys Ther. 2008 Apr;88(4):449-59. doi: 10.2522/ptj.20070251. Epub 2008 Jan 24. PMID 18218822
- [Result] Bjerk M, Brovold T, Skelton DA, Bergland A. A falls prevention programme to improve quality of life, physical function and falls efficacy in older people receiving home help services: study protocol for a randomised controlled trial. BMC Health Serv Res. 2017 Aug 14;17(1):559. doi: 10.1186/s12913-017-2516-5. PMID 28806904
- [Result] Bjerk M, Brovold T, Skelton DA, Bergland A. Associations between health-related quality of life, physical function and fear of falling in older fallers receiving home care. BMC Geriatr. 2018 Oct 22;18(1):253. doi: 10.1186/s12877-018-0945-6. PMID 30348098
- [Result] Bjerk M, Brovold T, Skelton DA, Liu-Ambrose T, Bergland A. Effects of a falls prevention exercise programme on health-related quality of life in older home care recipients: a randomised controlled trial. Age Ageing. 2019 Mar 1;48(2):213-219. doi: 10.1093/ageing/afy192. PMID 30615055
- [Result] Bjerk M, Brovold T, Davis JC, Skelton DA, Bergland A. Health-related quality of life in home care recipients after a falls prevention intervention: a 6-month follow-up. Eur J Public Health. 2020 Feb 1;30(1):64-69. doi: 10.1093/eurpub/ckz106. PMID 31169888
- [Result] Bjerk M, Brovold T, Davis JC, Bergland A. Evaluating a falls prevention intervention in older home care recipients: a comparison of SF-6D and EQ-5D. Qual Life Res. 2019 Dec;28(12):3187-3195. doi: 10.1007/s11136-019-02258-x. Epub 2019 Jul 30. PMID 31364036

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from February 2016 to February 2017. 865 older adults were assessed for eligibility. 320 had experienced a fall and received an invitation letter to participate in this study. Recruitment stopped when the sample size target (150) was expected to be reached.
Pre-assignment Details: 167 older adults consented to baseline testing. 12 did not met the inclusion criteria and were not considered enrolled in the study. 155 met the inclusion criteria and were randomized in either the intervention or control group.
Groups:
- Intervention: Exercise and education: Exercise according to the falls prevention programme. Information on motivation, the effectiveness of falls prevention and the importance of adherence.
- Control: Activities as usual.
Period: 3-months Follow-up
Arm/Group | Intervention | Control
Started | 77 | 78
Completed | 69 | 69
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Death | 1 | 2
Not completed — Missed first follow-up | 5 | 1
Period: 6-months Follow-up
Arm/Group | Intervention | Control
Started | 74 (5 subjects missed the first follow-up, but continued the study and were assessed at 6 months.) | 70 (1 subject missed the first follow-up, but continued the study and was assessed at 6 months.)
Completed | 71 | 64
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 77 | 78 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.1 (6.7) | 82.2 (6.7) | 82.7 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 62 | 123
  Male | 16 | 16 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Living alone [Count of Participants; unit: Participants] — If the participant is living alone, e.g. without a spouse or cohabitant.
  Participants | 64 | 67 | 131
Higher education [Count of Participants; unit: Participants] — Education exceeds 12 years in total.
  Participants | 25 | 31 | 56
Medications weekly [Mean (Standard Deviation); unit: medications] — No. of different medications, weekly
  medications | 5.1 (3.7) | 5.4 (3.2) | 5.3 (3.4)
Practical assistance [Count of Participants; unit: Participants] — Type of home care received
  Participants | 50 | 58 | 108
Nursing [Count of Participants; unit: Participants] — Type of home care received
  Participants | 20 | 27 | 47
Safety alarm service [Count of Participants; unit: Participants] — Type of home care received
  Participants | 61 | 56 | 117
Walking aid [Count of Participants; unit: Participants] — If a walking aid is used
  Participants | 60 | 54 | 114
Falls [Mean (Standard Deviation); unit: falls] — No. of falls in the last 12 months
  falls | 2.5 (3.3) | 2.9 (4.0) | 2.7 (3.7)
Falls injuries [Count of Participants; unit: Participants] — Minor injuries from falls in the last 12 months Population: One missing value
  Participants
    number analyzed (Participants) | 77 | 77 | 154
    No injuries | 17 | 13 | 30
    Minor injuries | 35 | 35 | 70
    Serious injuries, hospitalization | 25 | 29 | 54
Mini-Mental Statement Examination [Mean (Standard Deviation); unit: scores on a scale] — The Mini Mental Statement Examination (MMSE) is a measurement of global cognitive function. The highest score is 30, the lowest score is 0. A score below 23 indicates cognitive impairment which is an exclusion criteria in this study.
  scores on a scale | 27.4 (2.2) | 27.4 (2.2) | 27.4 (2.2)
Falls Efficacy Scale - International [Mean (Standard Deviation); unit: scores on a scale] — The Falls Efficacy Scale - International (FES-I) derives from a self-report questionnaire, assessing concerns about falling in 16 different daily activities. The total score ranges from 16 (no concern) to 64 (high concern).
  scores on a scale | 30.2 (10.1) | 31.1 (9.6) | 30.7 (9.8)
Instrumental Activities of Daily Living > 6 [Count of Participants; unit: Participants] — No. of participants with a score higher than 6 on the Instrumental Activities of Daily Living (IADL) scale, Lawton and Brody. It is a measure of a person's self-reported ability to perform complex activities of daily living. The summary score ranges from 0 (low function, dependent) to 8 (high function, independent).
  Participants | 42 | 45 | 87
Sit-to-stand test [Mean (Standard Deviation); unit: raises] — No. of raises from a chair in 30 seconds. From the sitting position, the subject stands completely up, then sits completely back down, repeated for 30 seconds.
  raises | 5.5 (3.8) | 4.7 (4.4) | 5.1 (4.1)
4-meter walk test [Mean (Standard Deviation); unit: m/s] — Population: One missing value
  m/s
    number analyzed (Participants) | 76 | 78 | 154
    (all) | 0.61 (0.18) | 0.63 (0.24) | 0.62 (0.21)
Berg Balance Scale [Mean (Standard Deviation); unit: scores on a scale] — The Berg Balance Scale is a 14-item scale, which is applied to assess static and dynamic balance in older adults. The summary score ranges from 0 (low, wheelchair bound) to 56 (high, independent)
  scores on a scale | 39.1 (11.1) | 39.1 (11.6) | 39.1 (11.3)
Mini Nutritional Assessment [Count of Participants; unit: Participants] — Risk of or being malnourished in the Mini Nutritional Assessment (MNA). The summary score of MNA ranges from 0 to 14, where a score below 12 indicates a risk of malnutrition or being malnourished.
  Participants
    No risk | 57 | 60 | 117
    Risk of or malnourished | 20 | 18 | 38
SF-36 Physical Component Summary [Mean (Standard Deviation); unit: scores on a scale] — Physical Component Summary in the Short Form 36 Health Survey (SF-36). SF-36 measures health-related quality of life. Its summary score is comprised of a physical component summary (PCS) and a mental component summary (MCS). The scores range from 0-100 (worst-best) in each scale.
  scores on a scale | 38.2 (9.0) | 38.4 (9.1) | 38.3 (9.0)
SF-36 Mental Component Summary [Mean (Standard Deviation); unit: scores on a scale] — Mental Component Summary in the Short Form 36 Health Survey (SF-36). SF-36 measures health-related quality of life. Its summary score is comprised of a physical component summary (PCS) and a mental component summary (MCS). The scores range from 0-100 (worst-best) in each scale.
  scores on a scale | 50.4 (9.9) | 48.4 (10.6) | 49.4 (10.3)
EQ-5D [Mean (Standard Deviation); unit: scores on a scale] — Health-related quality of life measured by the EuroQOL EQ-5D instrument. Preference weights for United Kingdom were employed to generate utility scores ranging from -0.59 to 1. A score of 1 is associated with a health state without problems.
  scores on a scale | 0.64 (0.21) | 0.60 (0.24) | 0.62 (0.23)

OUTCOME MEASURES:

1. Primary Outcome: Short Form 36 Health Survey Summary Scores
Description: Changes in the Short Form 36 Health Survey (SF-36) summary scores from baseline to 3-months follow-up. SF-36 measures health-related quality of life. Its summary score is comprised of a physical component summary (PCS) and a mental component summary (MCS). The scores range from 0-100 (worst-best) in each scale. A positive change in the summary score indicates a better health-related quality of life.
Time Frame: Baseline, 3 months, 6 months
Population: Intention-to-treat population. Multiple imputation using a predictive mean matching model with arm, age, sex and baseline values of the imputed variable as predictors.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 77 | 78
scores on a scale
  Change in PCS Baseline - 3-months follow-up | 3.7 (1.0) | -0.3 (0.9)
  Change in PCS Baseline - 6-months follow-up | 3.0 (0.9) | 0.1 (0.9)
  Change in MCS Baseline - 3-months follow-up | 0.7 (1.1) | 3.8 (1.2)
  Change in MCS Baseline - 6-months follow-up | 1.7 (1.1) | 4.7 (1.3)

2. Secondary Outcome: EQ-5D
Description: Changes in the EuroQOL EQ-5D instrument indicating changes in health-related quality of life. Preference weights for United Kingdom were employed to generate utility scores ranging from -0.59 to 1. A score of 1 is associated with a health state without problems. A positive change in EQ-5D indicates a better health-related quality of life.
Time Frame: Baseline, 3 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 77 | 78
scores on a scale
  3-months follow-up | 0.06 (0.02) | 0.005 (0.03)
  6-months follow-up | 0.11 (0.02) | -0.02 (0.03)

3. Secondary Outcome: Berg Balance Scale
Description: Changes in the Berg Balance Scale (BBS), a 14-item scale applied to assess static and dynamic balance in older adults. The summary score ranges from 0 (low, wheelchair bound) to 56 (high, independent)
Time Frame: Baseline, 3 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 77 | 78
scores on a scale
  Change Baseline - 3-months follow-up | 5.4 (0.8) | 3.1 (0.9)
  Change Baseline - 6-months follow-up | 4.9 (0.9) | 3.5 (0.9)

4. Secondary Outcome: Sit-to-stand Test
Description: Changes in the no. of raises in 30 seconds. From the sitting position, the subject stands completely up, then sits completely back down, repeated for 30 seconds.
Time Frame: Baseline, 3 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: raises
Arm/Group | Intervention | Control
Number analyzed (Participants) | 77 | 78
raises
  Change Baseline - 3-months follow-up | 1.2 (0.4) | 0.8 (0.4)
  Change Baseline - 6-months follow-up | 1.2 (0.4) | 1.1 (0.4)

5. Secondary Outcome: 4-meter Walk Test
Description: Changes in the 4-meter walk test. Participants are asked to walk a distance of 4 meters at their usual pace, measured in m/s
Time Frame: Baseline, 3 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Intervention | Control
Number analyzed (Participants) | 77 | 78
m/s
  Change Baseline - 3-months follow-up | 0.06 (0.02) | 0.06 (0.02)
  Change Baseline - 6-months follow-up | 0.05 (0.02) | 0.05 (0.02)

6. Secondary Outcome: Falls Efficacy Scale - International
Description: Changes in falls-efficacy measured with the Falls Efficacy Scale - International (FES-I) derives from a self-report questionnaire, assessing concerns about falling in 16 different daily activities. The total score ranges from 16 (no concern) to 64 (high concern). A decrease in scores indicates less concerns.
Time Frame: Baseline, 3 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 77 | 78
scores on a scale
  Change Baseline - 3-months follow-up | -1.7 (1.2) | -2.3 (1.1)
  Change Baseline - 6-months follow-up | -1.7 (1.2) | -1.3 (1.2)

7. Secondary Outcome: Instrumental Activities of Daily Living
Description: No. of participants with scores on the Instrumental Activities of Daily Living (IADL) scale, Lawton and Brody. IADL is a measure of a person's self-reported ability to perform complex activities of daily living. The summary score ranges from 0 (low function, dependent) to 8 (high function, independent).
Time Frame: Baseline, 3-months, 6-months
Population: Complete, non-missing observations for both groups at baseline. 69 participants completed the 3-months follow-up. In the intervention group, 71 participants completed the 6-months follow-up, with 1 missing observation on IADL. In the control group, 64 participants completed the 3-months follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 77 | 78
Participants
  Baseline: 0, low function | 0 | 0
  Baseline: 1 | 0 | 0
  Baseline: 2 | 0 | 1
  Baseline: 3 | 1 | 2
  Baseline: 4 | 7 | 7
  Baseline: 5 | 8 | 7
  Baseline: 6 | 19 | 16
  Baseline: 7 | 21 | 14
  Baseline: 8, high function | 21 | 31
  3-months follow-up: number analyzed (Participants) | 69 | 69
  3-months follow-up: 0, low function | 0 | 0
  3-months follow-up: 1 | 1 | 1
  3-months follow-up: 2 | 2 | 2
  3-months follow-up: 3 | 0 | 4
  3-months follow-up: 4 | 4 | 2
  3-months follow-up: 5 | 9 | 7
  3-months follow-up: 6 | 15 | 10
  3-months follow-up: 7 | 17 | 18
  3-months follow-up: 8, high function | 21 | 25
  6-months follow-up: number analyzed (Participants) | 70 | 64
  6-months follow-up: 0, low function | 0 | 1
  6-months follow-up: 1 | 2 | 1
  6-months follow-up: 2 | 1 | 4
  6-months follow-up: 3 | 3 | 3
  6-months follow-up: 4 | 2 | 6
  6-months follow-up: 5 | 9 | 7
  6-months follow-up: 6 | 9 | 9
  6-months follow-up: 7 | 20 | 8
  6-months follow-up: 8, high function | 24 | 25

8. Secondary Outcome: Walking Habits
Description: Questions regarding walking habits in the last 7 days. Summarized in total minutes walking.
Time Frame: Baseline, 3 months, 6 months
Population: At baseline, one observation was missing in the intervention group. 69 participants completed the 3-months follow-up. In the intervention group, 71 participants completed the 6-months follow-up. In the control group, 64 participants completed the 3-months follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 77 | 78
Participants
  Baseline: number analyzed (Participants) | 76 | 78
  Baseline: 0 min | 6 | 6
  Baseline: 0-30 min | 21 | 16
  Baseline: 30-90 min | 20 | 27
  Baseline: 90-180 min | 15 | 18
  Baseline: > 180 min | 14 | 11
  3-months follow-up: number analyzed (Participants) | 69 | 69
  3-months follow-up: 0 min | 9 | 17
  3-months follow-up: 0-30 min | 11 | 16
  3-months follow-up: 30-90 min | 16 | 16
  3-months follow-up: 90-180 min | 13 | 7
  3-months follow-up: > 180 min | 20 | 13
  6-months follow-up: number analyzed (Participants) | 71 | 64
  6-months follow-up: 0 min | 10 | 16
  6-months follow-up: 0-30 min | 15 | 13
  6-months follow-up: 30-90 min | 17 | 16
  6-months follow-up: 90-180 min | 13 | 8
  6-months follow-up: > 180 min | 16 | 11

9. Secondary Outcome: Mini Nutritional Assessment
Description: The summary score of the Mini Nutritional Assessment (MNA) maps to three nutritional statuses "Normal nutritional status", "Risk of malnutrition" and being "Malnourished".
Time Frame: Baseline, 3 months, 6 months
Population: Complete, non-missing observations for both groups at baseline. 69 participants completed the 3-months follow-up. In the intervention group, 71 participants completed the 6-months follow-up. In the control group, 64 participants completed the 3-months follow-up, but 3 observations are missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 77 | 78
Participants
  Baseline: Normal nutritional status | 57 | 60
  Baseline: At risk of malnutrition | 17 | 18
  Baseline: Malnourished | 3 | 0
  3-months follow-up: number analyzed (Participants) | 69 | 69
  3-months follow-up: Normal nutritional status | 48 | 44
  3-months follow-up: At risk of malnutrition | 21 | 21
  3-months follow-up: Malnourished | 0 | 4
  6-months follow-up: number analyzed (Participants) | 71 | 61
  6-months follow-up: Normal nutritional status | 55 | 35
  6-months follow-up: At risk of malnutrition | 14 | 23
  6-months follow-up: Malnourished | 2 | 3

10. Secondary Outcome: Exercise According to the Protocol. Adherence
Description: No. of participants in the intervention group performing exercises according to the protocol in the intervention period until 3-months follow-up. Participant are encouraged to complete an activity diary where they note if the exercise programme has been executed as planned. If they have not completed sufficient exercises, they are supposed to make a note in the diary.
Time Frame: Baseline and 3 months
Population: All subjects in the intervention group with nonmissing observations at 3-months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 68
Participants | 50

11. Secondary Outcome: No. of Participants Exercising Post-intervention
Description: Self-reported exercise behavior post-intervention between 3-months follow-up to 6-months follow-up.
Time Frame: 3 months and 6 months
Population: All subjects with nonmissing observations at 6-months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 71 | 63
Participants
  None | 14 | 23
  Individual exercise | 46 | 25
  Group exercise | 3 | 11
  Both | 8 | 4

12. Secondary Outcome: No. of Falls
Description: No. of falls in the post-intervention period between 3-months follow-up and 6-months follow-up. Falls are defined as an event, i.e. fall, trip, slip, which results in the person coming to rest on the ground or floor or other lower level.
Time Frame: 3 months and 6 months
Population: All subjects with nonmissing observations at 6-months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 71 | 64
Participants
  No falls | 57 | 41
  One or more falls | 14 | 23

ADVERSE EVENTS:
Time Frame: Study period of 6 months
Description: Adverse events definition also included falls, cardiovascular events or musculoskeletal injuries when performing exercises.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 3/77 | 3/78
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/78
Other Adverse Events (participants affected / at risk) | 3/77 | 0/78
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=77) | Control (N=78)
Musculoskeletal pain/discomfort (Musculoskeletal and connective tissue disorders) | 3 | 0 — Musculoskeletal pain/discomfort after using ankle cuffs

LIMITATIONS AND CAVEATS:
Some measurements are self-reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT02374307/Prot_SAP_000.pdf